CLINICAL TRIAL: NCT03222362
Title: Pars Plana Vitrecromy in Patients Aged 85 Years and Above
Acronym: PPV
Status: Completed | Type: Observational
Sponsor: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, Adiel Barak, Head Of vitrerretinal service, Tel Aviv Medical Center
Other Study IDs: 0542-15-TLV
Record Dates: First submitted 2017-07-16; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Vitreous Injury; Retinal Detachment; Age Related Macular Degeneration
Keywords: retinal detachment; trauma; age related macular degeneration
MeSH Terms: conditions — Retinal Detachment; Macular Degeneration; Wounds and Injuries | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients 85 years and above: 120 consecutive patients (male and female), aged 85 years and above, who underwent pars plana vitrecromy in the Tel Aviv Medical Center during the years 01/01/2006 - 31/12/2013, and were followed by physicians in the ophthalmology department in the center until December 2015.
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery

SUMMARY:
We reviewed the records of 120 consecutive patients (male and female), aged 85 years and above, who underwent pars plana vitrecromy in the Tel Aviv Medical Center during the years 01/01/2006 - 31/12/2013, and were followed by physicians in the ophthalmology department in the center until December 2015.

DETAILED DESCRIPTION:
We reviewed the records of 120 consecutive patients (male and female), aged 85 years and above, who underwent pars plana vitrecromy in the Tel Aviv Medical Center during the years 01/01/2006 - 31/12/2013, and were followed by physicians in the ophthalmology department in the center until December 2015. We will be measuring visual acuity, intra-ocular pressure, demographics (age, gender), indication for surgery, ocular co-morbidities, surgical parameters (time of surgery, type of anesthesia - general or local, type of suture), and intraoperative and postoperative complications.

Primary outcome - visual acuity will be measured at base line, after 1 week, 1 month, 3 months, 6 months / last follow up (until December 2015). visual acuity will be determined by a standardized chart test (Snellen chart). For statistical analysis, all VA values were converted to logMAR scale. According to Holladay and the University of Freiburg study group results, blindness was set at 0.00125/2.9 (decimal/logMAR), light perception at 0.0025/2.6, hand movements at 0.005/2.3 and counting fingers at 0.014/1.85. Data will be analyzed using SPSS software. A p-value of 0.05 will be considered statistically significant and t-tests analysis will be used to compare between means.

Secondary outcomes - demographics, Indication for surgery, ocular co morbidities will be measured at baseline. Surgical parameters and intraoperative complications will be measured at 1 week. Postoperative complications will be measured during follow up after 1 week, 1 month, 3 months, 6 months / last follow up (until December 2015).

Complications will be measured by examination of intraocular pressure, slit-lamp and fundus (Ophthalmoscopic Exam).

ELIGIBILITY:
Inclusion Criteria:

Patients aged 85 years and above, who underwent pars plana vitrecromy in the Tel Aviv Medical Center during the years 01/01/2006 - 31/12/2013

Exclusion Criteria:

ANy other

Min Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 85 years and above, who underwent pars plana vitrecromy in the Tel Aviv Medical Center during the years 01/01/2006 - 31/12/2013
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
visual acuity | study entry until December 2015 .
  visual acuity in Snellen chart

SECONDARY OUTCOMES:
Postoperative complications | study entry until December 2015 .
  Postoperative complications will be measured during follow up after 1 week, 1 month, 3 months, 6 months / last follow up